CLINICAL TRIAL: NCT06670729
Title: Psychotherapeutic Effect of Listening to Quran Recitation on Dental Anxiety: a Randomized Controlled Trial
Brief Title: Alternatives to Manage Dental Fear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Abrar Nizar Al-Attar, assistant lecturer, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: REC108
Record Dates: First submitted 2024-10-30; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Fear Anxiety; Discomfort; Psychotherapy Intervention Evaluation
Keywords: Quran; fear; discomfort; dentistry

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The dentist who provides dental care was blinded to the assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Quran listening group (Experimental): participants listen to Quran recitation
  Interventions: Other: Quran listening
- silent headphones (Other): participant's headphone is silent
  Interventions: Other: silent headphones group

INTERVENTIONS:
Other: Quran listening — listening to quran recitation via head phone
  Arms: Quran listening group
Other: silent headphones group — headphones were silent, patient do not listen to any thing
  Arms: silent headphones

SUMMARY:
This study compares the psychological effects on patients attend the dental clinic by listening to specific audios

DETAILED DESCRIPTION:
Participants of the experimental group listened to Quran recitation using auto-controlled headphones, whereas headphones of the control group participants were silent then the two groups answer questionnaire prepared for this purpose.

ELIGIBILITY:
Inclusion Criteria:

* any patient eligible for dental treatment
* willing to participate

Exclusion Criteria: participants

* less than 18 years of age,
* mentally retarded,
* had hearing impairment or deafness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
fear | before, during and immediately after dental session
  fear was assessed using a questionnaire that is based on Dental anxiety scale (DAS) and Modified Dental Anxiety scale (MDAS), statistically significant descending ranks of fear reflects effectiveness of the intervention, when statistical analysis was significant, clinical (practical) effect size was also obtained to determine the clinically effective modality of management
discomfort | during and immediately after dental session
  presence or absence of discomfort was assessed using dental anxiety scale and modified dental anxiety scale, descending ranks of fear reflects effectiveness of the intervention

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No